CLINICAL TRIAL: NCT00679068
Title: Effects of 12 Weeks Treatment With Bosentan on Respiratory Mechanics in Patients With Pulmonary Hypertension
Brief Title: Effects of Bosentan on Respiratory Mechanics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment of patients
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief ICU, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 525FSM
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Hypertension
Keywords: respiratory mechanics; bosentan; exercise capacity
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): treatment with Bosentan
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — 62.5 mg b.i.d. for 4 weeks, then 125 mg b.i.d.for the remaining 8 weeks (if tolerated)

SUMMARY:
Bosentan has been largely used in the treatment of pulmonary hypertension (PH). It can improve exercise capacity, lower Borg dyspnoea score nad these effects are usually associated with the concomitant improvement in cardiopulmonary haemodynamics.

No physiological study has so far verified the hypothesis that Bosentan may laso have an effect on the "respiratory side" of the cadio-pulmonary system (i.e. on pulmonary mechanics and work of breathing)

DETAILED DESCRIPTION:
Endothelins are powerful vasoconstrictor peptides that also play numerous other functions in many different organs. Endothelin-1 (ET-1) is the most abundant and important of this family of peptides in blood vessels. Production of ET-1 is increased in the endothelium and the kidney in salt-dependent models of hypertension ET-1 elicits an inflammatory response by increasing oxidant stress in the vascular wall, which induces vascular remodeling and endothelial dysfunction found in the hypertensive models that exhibit an endothelin-mediated component. Endothelin receptor antagonists lower blood pressure in hypertensive patients. They could become therapeutic agents for prevention of target organ damage in hypertension and in type 2 diabetes, chronic renal failure and congestive heart failure. Side effects of endothelin receptor blockers have prevented up to the present their development for these indications. Endothelin antagonists have been approved only for the treatment of pulmonary hypertension, a rapidly fatal condition in which the endothelin system plays an important role and endothelin antagonists exert favorable effects.The exact mechanism of action of ERAs on the pulmonary vascular bed remains unclear. Vasodilatation is just a part of the mechanism, since usually 70%-80% of Idiopathic PAH patients do not respond acutely to vasodilators. Endothelin is likely to be involved in pulmonary vasoconstriction, inflammation, cellular proliferation and fibrosis ie. remodelling Recent research illustrates that bosentan is capable of blunting the vascular remodelling normally associated with PAH If ERAs could prevent remodelling, they might substantially improve the long-term survival in patients with mild symptoms (WHO class II or I).

Bosentan, the most popular endothelin receptor antagonist, has been largely used in the treatment of pulmonary hypertension (PH). It can improve exercise capacity, lower Borg dyspnoea score nad these effects are usually associated with the concomitant improvement in cardiopulmonary haemodynamics.

No physiological study has so far verified the hypothesis that Bosentan may laso have an effect on the "respiratory side" of the cadio-pulmonary system (i.e. on pulmonary mechanics and work of breathing)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with World Health Organization (WHO) functional class II-III.
* A systemic pulse oximetry (SpO2) between 70% and 90% at rest with room air and a baseline 6-minute walk distance between 150 and 450 m were required for inclusion.
* PAH confirmed by cardiac catheterization as mean pulmonary arterial pressure greater or equal to25 mm Hg, pulmonary capillary wedge pressure lower 15 mm Hg,

Exclusion Criteria:

* Patients were excluded if they had patent ductus arteriosus (for hemodynamic assessment difficulties)
* complex congenital heart defect
* left ventricular dysfunction (left ventricular ejection fraction lower 40%)
* restrictive lung disease (total lung capacity lower 70% predicted)
* obstructive lung disease (forced expiratory volume in 1 second [FEV1] lower 70% predicted
* with FEV1/forced vital capacity lower 60%)
* or previously diagnosed coronary artery disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics (i.e. lung compliance, resistances and work of breathing) | 12 weeks

SECONDARY OUTCOMES:
exercise capacity (i.e. 6 mwd), dyspnea, oxygen saturation and cardiac function (i.e. hemodynamic evaluation) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, Principal Investigator — Fondazione S.Maugeri
Locations (1):
- Respiratory Unit, Fondazione S.Maugeri, Pavia, PV, Italy